CLINICAL TRIAL: NCT06567275
Title: Analgesic Effect of Ultrasound Guided Erector Spinae Plane Block Versus Serratus Anterior Plane Block in Pediatric Patients Undergoing Aortic Coarctectomy , a Randomized Controlled Study .
Brief Title: Comparison Between Serratus Anterior Plane Block and Erector Spinae Plane Block in Coarctectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Awad Eissa Roman, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Nerve blocks in coarctectomy
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-08

CONDITIONS: Aortic Coarctation
Keywords: erector spinae plane block; serratus anterior plane block; aortic coarctectomy
MeSH Terms: conditions — Aortic Coarctation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erector spinae plane block (Experimental): Ultrasound-guided erector spinae plane block will be done by injecting 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%).
  Interventions: Procedure: Erector Spinae Plane Block
- serratus anterior plane block (Experimental): Ultrasound-guided serratus anterior plane block will be done by injecting 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%).
  Interventions: Procedure: Serratus Anterior Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Ultrasound-guided erector spinae plane block will be done by injecting 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%)
  Arms: erector spinae plane block
Procedure: Serratus Anterior Plane Block — Ultrasound-guided serratus anterior plane block will be done by injecting 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%)
  Arms: serratus anterior plane block

SUMMARY:
Pain is considered to be subjective, however, in children, it is believed to be felt rather than expressed because they often depend on the caregiver for their safety and well-being.

There is significant pain after thoracotomy surgery because of pleural and muscular damage, ribcage disruption, and intercostal nerve damage during surgery, which if not effectively managed, will lead to various systemic complications; pulmonary (atelectasis, pneumonia, and stasis of bronchial secretions), cardiovascular (increased oxygen consumption and tachycardia), musculoskeletal (muscle weakness), increased neurohormonal response and prolonged hospital stay. So adequate and sufficient post-operative analgesia for pediatric patients is mandatory.

The use of highly potent opioids for pediatric cardiothoracic anesthesia has gained widespread popularity during the last 20 years. In addition to the important advantage of hemodynamic stability, the large-dose opioid-based anesthetic techniques also blunt the stress response, However, large doses can cause oversedation, respiratory depression, and prolonged mechanical ventilation after surgery.

serratus anterior plane block guided by ultrasound was developed by Blanco et al, it is a novel technique in the management of pain following thoracic procedures.

Local anesthetic inserted into these planes will spread throughout the lateral chest wall, resulting in paresthesia of the T2 through T9 dermatomes of the anterolateral thorax. It became popular because it is much safer and easily administered than other alternative regional techniques such as thoracic paravertebral and thoracic epidural blocks.

The Erector Spinae Plane Block (ESPB) is also one of the recently known pain-controlling techniques used in pediatric cardiothoracic surgeries. It became popular because it is much safer and easily administered than other alternative regional techniques such as thoracic paravertebral and thoracic epidural blocks. Chin et al. documented the cadaveric spread of local anesthetic and noted that, radiologically, the local anesthetic spread extended 3 or 4 levels cranially and caudally from the site of injection.

These two blocks have been compared in a study by wang HJ et al in patients undergoing radical mastectomy.

To our knowledge, the comparison of serratus Plane Block versus erector spinae plane block in aortic coarctectomy operations in pediatric patients has not been investigated yet. This has encouraged the performance of the present study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3 months-2 years.
* RACHS-1 score 3.
* Patients undergoing aortic coarctectomy operation with Lateral thoracotomy incision.

Exclusion Criteria:

* Patients whose parents or legal guardians refuse to participate.
* Preoperative mechanical ventilation.
* Preoperative inotropic drug infusion.
* Perioperative cardiopulmonary arrested patients.
* Patients undergoing aortic coarctectomy operation with midline sternotomy incision.
* History of mental retardation or delayed development that may interfere with pain intensity assessment.
* Known or suspected coagulopathy. (PT < 75% of control)
* Any congenital anomalies or any infection at the site of injection.
* Known or suspected allergy to any of the studied drugs.
* liver enzymes elevated more than the normal values.
* Renal function impairment (Creatinine value more than 1.2mg/dl or BUN more than 20mg/dl).
* Heart failure patients
* Redo patients and previous catheter dilatations

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2024-08-24 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Total intraoperative fentanyl consumption by mcg/kg. | Intra-operatively up to extubation
  calculating the total dose of fentanyl used intraoperatively

SECONDARY OUTCOMES:
Time (in minutes) to 1st rescue analgesia (morphine) | 1st 24 hours postoperatively
  estimating the time of the need for 1st dose of morphine which was given for pain scores ≥ 4
Heart rate and systolic blood pressure | up to 15 minutes after extubation
  recorded at 5 minutes after intubation (baseline value), before skin incision at 15 minutes after the block, after skin incision, after rib retraction, after aortic clamping, after aortic declamping, immediately after skin closure, and at 15 minutes after extubation
The need and the dose of sodium nitroprusside after aortic clamping | from aortic clamping until removal of the clamps
  sodium nitroprusside was given to control the hypertensive response to aortic clamping
total morphine dose | up to 24 hours after surgery
  morphine was given for pain scores ≥ 4
Face, Legs, Activity, Cry, Consolability (FLACC) score | up to 24 hours after surgery
  Postoperative pain was assessed using the Face, Legs, Activity, Cry, Consolability (FLACC) score every 2 hours for the first 24 hours postoperatively. If the FLACC score ≥ 4, 0.02 mg/kg morphine IV was administered as rescue analgesia to be repeated every 15-20 minutes till the pain score reaches < 4, not exceeding 0.2 mg/kg every 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa M Elsadeq, Study Director — Professor of Anesthesia, Pain Management, and Surgical ICU Faculty
Locations (1):
- Abu Elreish Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gado AAM, Atia MAM, Roman AA, Elsadeq WM, Jaccoub VF. Analgesic efficacy of ultrasound guided erector spinae plane block versus serratus anterior plane block in pediatric patients undergoing aortic coarctectomy; a randomized controlled study. BMC Anesthesiol. 2025 Jul 30;25(1):370. doi: 10.1186/s12871-025-03256-y. PMID 40739624